CLINICAL TRIAL: NCT04568564
Title: Telerehabilitation of Reduced Physiotherapy Service in SARS-CoV-2 Pandemic Process in Lung Surgery Patients
Brief Title: Telerehabilitation in Lung Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PostopTele
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer; Physiotherapy
Keywords: exercise; videoconference; lung cancer; surgery; postoperative; chest physiotherapy; telerehabilitation
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Breathing Exercises; Walking

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Group (TG) (Experimental): Patients diagnosed with lung cancer and underwent thoracotomy
  Interventions: Other: Breathing exercise, intensive spirometry use, supported cough, progressive mobilisation and ambulation
- Control group (CG) (Active Comparator): Patients diagnosed with lung cancer and underwent thoracotomy
  Interventions: Other: Exercise booklet

INTERVENTIONS:
Other: Breathing exercise, intensive spirometry use, supported cough, progressive mobilisation and ambulation — The exercise program includes breathing exercises (chest-abdominal-lateral basal breathing; 10 repetitions), use of intensive spirometry (20 repetitions) and assisted coughing. Apart from this, a progressive mobilization program will be applied considering patient tolerance and hemodynamic parameters, starting after the patient is taken to the service room. The teleconference exercise call will be continued from the postop 1st day until discharge, twice a day.
  Arms: Telerehabilitation Group (TG)
Other: Exercise booklet — Patients will be interviewed by videoconferencing method at least 1 day before the operation, their first evaluation will be taken and an exercise booklet will be given.
  Arms: Control group (CG)

SUMMARY:
In this study, providing access to physiotherapy applications by telerehabilitation method and the effectiveness of this application will be examined for patients who have undergone lung surgery in the early postoperative period during the pandemic process in which social isolation continues.

DETAILED DESCRIPTION:
* Patients who meet the inclusion criteria and agree to participate in the study will be included in the study.
* Patients diagnosed with lung cancer and underwent thoracotomy will be randomly divided into Telerehabilitation Group (TGR) and Control (KG) groups.
* Before the operation, enlightened and signed consent will be obtained from the cases, the first evaluations of the patients in both groups will be made and the first exercise training will be given to the telerehabilitation group.
* The study group will be followed up every day during their hospitalizations and the final tests of both groups will be made before discharge. Long-term follow-up will be carried out in the 1st month and 3rd month after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Having a smart phone and capable of making video calls,
* Planned to be operated with thoracotomy or videothoracoscope,
* Staged between IA and IIIB with clinical staging,
* With proven lung tumor (If AC diagnosis is not confirmed after frozen or wedge, the patient will be excluded from the study),
* Patients with no cardiac disease (ASA II or better) that affects their quality of life.

Exclusion Criteria:

* Having a cardiac disease that affects the quality of life,
* Serious cognitive problems and presence of psychiatric diseases,
* Presence of physical limitations (vision, hearing impairment, orthopedic problems).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Major complication rate | Up to 3 months
  Major complication rates such as postoperative fever, infection, and hemorrhage will be documented.

SECONDARY OUTCOMES:
The six-minute walking test | Up to 3 months
  The six-minute walking test is an example of timed distance testing, widely used in clinical research and rehabilitation studies. According to the guidelines published by the American Thoracic Society, 6MWT is an easy-to-use, better tolerated test that reflects daily activities better than other walking tests. It can be applied in a short time. Requires little equipment. The six-minute walk test, used as a field test, is a simple and inexpensive test compatible with daily activities, which does not require exercise equipment. Before starting the test, the patient should rest for at least 10 minutes by sitting in the chair near the starting point. The walking area must be at least 30 m long. A shorter corridor causes more time to be spent for more frequent turns and changes of direction. With the help of stopwatch, it is kept for 6 minutes and the number of laps during the period is calculated and recorded. The functional capacity of the cases will be evaluated with 6MWT.
Modified Medical Research Council Dyspnea Scale | Up to 3 months
  It is a scale used to determine the severity of dyspnea with a rating of zero to 4. Zero means no dyspnea perception and 4 means severe dyspnea.
Visual analog scale | Up to 3 months
  The pain, dyspnea and fatigue level of the cases were evaluated with visual analog scale (VAS) score. The scale presented as a 100 mm horizontal ruler is a documented method for scoring continuous soft data. "0" score means no pain, "100" means very severe pain
Duration of tube thoracostomy drainage | Up to 3 months
Forced expiratory volume one second (FEV1) | Up to 3 months
  FEV1 measurements will be reported as absolute values (e.g. liters, measured) and percentage of predicted (FEV1measured/ FEV1 predicted).
Forced vital capacity (FVC) | Up to 3 months
  FVC measurements will be reported as absolute values (e.g. liters, measured) and percentage of predicted (FVCmeasured/ FVC predicted).
Diffusion Capacity | Change from baseline to 1 and 3 months
  DLCO and DLCO / VA values will be analyzed
Lung Capacities | Change from baseline to 1 and 3 months
  Lung capacities will be given the measured value and their percentages will be calculated according to the estimated values.
Lung V/Q Scintigraphy | Change from baseline to 1 and 3 months
  Tumor side and contralateral lung V / Q scintigraphy measurements will be made.
Procalcitonin (PCT) | Up to 3 months
  Procalcitonin is a substance produced by many types of cells in the body, often in response to bacterial infections but also in response to tissue injury. The level of procalcitonin in the blood can increase significantly in systemic bacterial infections and sepsis.The reference value of PCT in adults and children older than 72 hours is 0. 15 ng/mL or less.
C-Reactive Protein (CRP) | Up to 3 months
  C-reactive protein is a substance produced by the liver in response to inflammation. For a standard CRP test, a normal reading is less than 10 milligram per liter (mg/L). A test result showing a CRP level greater than 10 mg/L is a sign of serious infection, trauma or chronic disease, which likely will require further testing to determine the cause
Ferritin | Up to 3 months
  Ferritin is a blood protein that contains iron. The normal ferritin levels range from 12 to 300 nanograms per milliliter of blood (ng/mL) for males and 12 to 150 ng/mL for females.
Lactate dehydrogenase | Up to 3 months
  Lactate dehydrogenase is an enzyme that helps turn sugar into energy for your cells. High LDH levels could indicate cell damage.Normal LDH levels range from 140 units per liter (U/L) to 280 U/L or 2.34 microkatals/L to 4.68 microkatals/L.
D'dimer test | Up to 3 months
  D-dimer tests are used to help rule out the presence of an inappropriate blood clot (thrombus). The reference concentration of D-dimer is < 250 ng/mL, or < 0.4 mcg/mL.
Partial Carbon monoxide Pressure (PaCO2) | Up to 3 months
  The partial pressure of carbon dioxide (PCO2) is the measure of carbon dioxide within arterial or venous blood. It often serves as a marker of sufficient alveolar ventilation within the lungs. Generally, under normal physiologic conditions, the value of PCO2 ranges between 35 to 45 mmHg.
Partial Oxigen Pressure (PaO2) | Up to 3 months
  The partial pressure of oxygen, also known as PaO2, is a measurement of oxygen pressure in arterial blood. 75 to 100 millimeters of mercury (mm Hg) is the normal ranges.
Arterial blood oxygen saturation level (SaO2) | Up to 3 months
  It reflects the saturation level of hemoglobin with oxygen. Its normal values are 95-100%.
Anxiety inventory | Up to 3 months
  The state-trait anxiety scale will determine the anxiety levels of patients before and after surgery. It is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic.While evaluating, a score between 1 (or -1) and 4 (or -4) is given for each item according to the positive or negative characteristics of the item, and the total score to be obtained is 50 constant is added. The highest score is 80, the lowest is 20. Total anxiety the higher the score, the more anxiety level of the person filling the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine Thoracic Surgery Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided